CLINICAL TRIAL: NCT04675840
Title: Intrathecal Morphine for Robotic-assisted Laparoscopic Hysterectomy- a Prospective Randomized Controlled Study.
Brief Title: Intrathecal Morphine for Robotic-assisted Laparoscopic Hysterectomy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karlstad Central Hospital (Other)
Responsible Party: Principal Investigator, Ragnar Henningsson, Associate Professor, Karlstad Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KarlstadCH
Record Dates: First submitted 2020-11-11; First posted 2020-12-19 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intrathecal morphine (Active Comparator): Spinal injection of 15mg Bupivakain and 0,25mg morphine before surgery.
  Interventions: Procedure: Robotic-assisted hysterectomy
- opiate po/iv (Active Comparator): Patient given 10mg Oxycodone orally before surgery.
  Interventions: Procedure: Robotic-assisted hysterectomy

INTERVENTIONS:
Procedure: Robotic-assisted hysterectomy — Robotic-assisted surgery

SUMMARY:
Is there any difference in the intensity of postoperative pain, nausea, urinary retention and legth of hospital stay in patients undergoing robotic assisted laparoscopic surgery if they receive intrathecal morphine or peroral and intravenous opiates during the surgery and is there a significant difference in the need of opiates after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients accepted for robotic-assisted laparoscopic surgery

Exclusion Criteria:

* Coagulopathy,
* Prior spine surgery,
* Chronic pain problems,
* Drug abuse,
* Pregnancy
* < 18 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Hysterectomy
Enrollment: 100 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Postop morphine consumption | First 48 hours after surgery
  Amount of opiates given postop
Postop grade of nausea & vomiting | First 24 hours after surgery
  Amount of antemetics given

SECONDARY OUTCOMES:
Hospital length of stay. | Up to 7 days
  Time from surgery (day 0) until Fit For Discharge FFD, defined as: 1) is taking oral pain medication only; 2) is able to walk around independently; 3) is tolerating full oral diet and have bowel movements; 4) is hemodynamically an respiratory stable; 5) has no drains or urinary catheter.
Patient overall satisfaction score. | Up to 7 days.
  1-10, where 1 is unsatisfied and 10 is very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Ragnar N Henningsson, Associate Professor, Principal Investigator — Dpt of Anesthesiology & Intensive Care
Locations (1):
- Department of Anesthesia & Intensive Care, Karlstad, Värmland County, Sweden

REFERENCES:
- [Derived] Engstrom AJE, Ivarsson CA, Aldergard A, Henningsson RN. Analgesic effects of intrathecal morphine and bupivacaine during robotic-assisted surgery: A prospective randomized controlled study. Pain Pract. 2023 Jul;23(6):631-638. doi: 10.1111/papr.13233. Epub 2023 Apr 18. PMID 37073442